CLINICAL TRIAL: NCT03015818
Title: Assessment of Osteoblastic Activity With 18F-Fluoride in Aortic Bioprosthesis Structural Valve Dysfunction (SVD)
Acronym: TEP-SVD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC16_0137
Record Dates: First submitted 2017-01-02; First posted 2017-01-10 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aortic Bioprosthesis Structural Valve Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Fluoride PET-CT ; CT calcium scoring ; 18F-FDG PET-CT (Experimental)
  Interventions: Other: 18F-Fluoride PET-CT ; CT calcium scoring ; 18F-FDG PET-CT

INTERVENTIONS:
Other: 18F-Fluoride PET-CT ; CT calcium scoring ; 18F-FDG PET-CT — 18F-Fluoride PET-CT CT calcium scoring 18F-FDG PET-CT

SUMMARY:
Structural valve dysfunction (SVD) is the most common and life threatening complication in patients treated by aortic valve replacement. A calcification process is frequently involved in SVD but its pathophysiology remains unclear. In the hypothesis of an active metabolic phenomenon of calcification, as previously shown in native aortic valve stenosis, rather than a passive deposit of calcium in valve tissue, positon emission tomography (PET) imaging with 18F-Fluoride could emphasize increased osteoblastic activity in SVD tissue.

This study will include patients with echocardiography-confirmed SVD. Echocardiographic parameters and other current parameters analyzed in SVD patients such as bioprosthesis calcium scoring derived from CT will be compared to 18F-Fluoride activity.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* written informed consent
* SVD defined on echocardiography by an alteration of bioprosthesis leaflets function with a mean transvalvular gradient > 20 mmHg and maximal velocity ≥ 3 m/s and effective orifice area ≤1.2 cm², and/or an aortic regurgitation more or equal to grade 2 on 4.

Exclusion Criteria:

* Inability to give informed consent
* Pregnancy
* Concurrent antibiotherapy
* Certain infectious endocarditis
* Concurrent anti-inflammatory therapy, including corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
18F-Fluoride activity | The day of the inclusion
  18F-Fluoride activity in valvular tissue will be determined by a tissue to bloodpool ratio of SUV (TBR). Patients will be divided in two groups : moderate SVD (EOA ≥ 0.8 and ≤ 1.2 cm²), and severe SVD (EOA ≤ 0.8 cm²), and TBR will be compared between the two groups, determined at time of inclusion.

SECONDARY OUTCOMES:
TBR in 18F-FDG | 6 months
  TBR in 18F-FDG will be compared between the two groups to analyze the inflammatory activity part in the SVD process
Both 18F-Fluoride and 18F-FDG TBR correlation | 6 months
  Both 18F-Fluoride and 18F-FDG TBR will be correlated with bioprosthesis calcium scoring and the following echocardiographic bioprosthesis function parameters : aortic regurgitation grade (none, trace, mild, moderate, severe) ; trans-valvular maximal velocity (m/s) ; mean trans-valvular gradient (mm Hg) ; EOA (cm²) ; visual echographic degenerescence score.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France